CLINICAL TRIAL: NCT03131804
Title: Effect of Intradialytic Exercise Among Hemodialysis Patients in the United Arab Emirates on Cardio-Metabolic Markers, Dialysis Adequacy, Quality of Life and Cost Effectiveness
Brief Title: Effect of Intradialytic Exercise In The United Arab Emirates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zayed University (Other)
Responsible Party: Principal Investigator, Mirey Karavetian, Assistant Professor, Zayed University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9637
Record Dates: First submitted 2017-04-17; First posted 2017-04-27 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Exercise; Dialysis
Keywords: Aerobic; Intradialytic; Cardio-metabolic markers; Dialysis Adequacy; Quality of Life; Cost Effectiveness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Participants (Experimental): Patients will represent their own controls (pre and post intervention), in the HD unit of Al Qassimi Hospital, Sharjah, United Arab Emirates.
  Interventions: Other: Intradialytic aerobic low intensity exercise

INTERVENTIONS:
Other: Intradialytic aerobic low intensity exercise — Intradialytic aerobic low intensity exercise program of 45 minutes per each hemodialysis session throughout the 6-month study duration

SUMMARY:
Hemodialysis (HD) patients have decreased physical functioning, diminished muscle mass and altered muscle quality thus the increased mortality rate compared to their age-matched population. Risk factors include their sedentary lifestyle and altered nutritional status [1]; the sedentary lifestyle or the lack of exercise is known to be a risk factor for cardiovascular complications [2] and contributes to worsen protein energy wasting (PEW), which is described as the loss of body protein mass and fuel reserves [1]. Therefore the health of the HD patients and consequently their quality of life (QOL) is deteriorated.

Studies have shown that aerobic exercise during HD improves aerobic capacity, blood pressure, heart rate, muscular strength, dialysis efficacy and quality of life; however, such studies were not done on the United Arab Emirates (UAE) HD patients and there is no protocol for implementing exercise in the UAE HD units [3-4]

Hypothesis: Intradialytic aerobic exercise will result in significantly improved clinical, cardio-metabolic and quality of life outcomes and reduced cost of care.

Primary objective of the study:

- To investigate whether the intradialytic exercise (IDE) within the routine practice of hemodialysis in the UAE will improve adequacy of dialysis.

Secondary objectives of the study:

* To study the effect of clinical and cardio-metabolic outcomes of the HD patients.
* Explore whether the trial would improve the cost effectiveness of this patient population's health care
* Define the nature of the IDE programs (intensity, duration, modality), and feasibility of its application in routine setting.

Importance of this research:

* Pioneering research in the Middle East and Gulf Cooperation Council (GCC) countries where the effect of intradialytic exercise will be studied for the first time on Arab population.
* It will contribute in identifying the exact strategies to integrate within the hemodialysis unit to improve clinical and cardio-metabolic outcomes, quality of life and healthcare cost.

Usefulness of this research to the UAE

* It will improve the health care cost and reduce cost wastage in the UAE (lean management).
* It will put UAE on the pedestal in front of other countries in integrating innovative methods for a better care of hemodialysis patients.

DETAILED DESCRIPTION:
Each patient will be asked to follow an Intradialytic aerobic low intensity exercise program of 45 minutes per each HD session throughout the 6-month study duration. The exercise will be tailored to each HD patient's ability (measured by VO2Max), supervised by the hospital physiotherapist and the research team. Continuous support and encouragement to the patients will be provided to assure they complete the 45 minutes of exercise on each HD session. Additionally, patients will be educated on the health benefits of exercise and how to integrate safe exercise into their daily life (by the research assistants).

Research assistants will be trained by the principal investigator (PI) on the study instruments and data collection methods. These assistants will administer 4 questionnaires (5 minutes each) for each HD patient separately and will collect data from the medical chart of each patient. The assessment will take place during the HD session.

The research assistants will also collect from the patient's file blood test results on a monthly basis (relevant to the study mentioned in table1); additional needed parameters will be analysed from the same blood sample that the hospital already collect for the patients monitoring, and will be analysed by the hospital for a fee from the research fund. For the β-aminoisobutyric acid (BAIBA) tests - cardiometabolic marker, 5 ML of the blood sample from each patient will be transported to a specialized lab for analysis.

All of the parameters, except the demographics (collected only at t0), will be collected and monitored at 3 time points: Baseline (t0), post-intervention (t1) and follow up (t2).

Assessment tools include

* Demographics: Height - Weight - Age - Social and Work status - Comorbidities - Education level
* Biochemical markers: C-reactive protein, Urea reduction ration, Phosphorus (P), BAIBA, Vitamin D3, Parathyroid Hormone, Calcium and Phosphorus Product
* Number of hospitalization days and emergency HD sessions
* Exercise Behavior questionnaire consists of 7 questions to assess the activity level of the patient before implementing the program. It will reflect the patient's activity level and importance.
* Barriers to physical activity questionnaire [5], which includes questions related to different categories of disease- and patient- specific barriers to physical activity (psychological, physical, and economical barriers) in addition to the lack of time factor.
* Malnutrition Inflammation Score (MIS) [6]: This is a comprehensive scoring system with significant associations with prospective hospitalization and mortality as well as measures of nutrition, inflammation, and anemia in HD. MIS has 10 components, each with four levels of severity from 0 (normal) to 3 (severely abnormal). The sum of all 10 MIS components ranges from 0 (normal) to 30 (severely abnormal); a higher score reflects more severe degree of malnutrition and inflammation. The scoring sheet consists of four sections.
* Quality of life (QOL) measured using the EuroQOL -5 health questionnaire [7]. It assesses 5 health concepts: mobility, self-care, usual activities (work, study, housework, and family or leisure activities), pain / discomfort, and anxiety / depression. Patients have 5 choices for each question to choose from to describe their health today. In addition, patients have to indicate on a scale marked from 0-100 their opinion about how good or bad their health state is today.
* Exercise effort test: Heart rate monitoring to assess the level of exercise performed [8]
* Exercise Fitness Level: measure using the Borg Scale of perceived Exertion [9]

All questionnaires that are originally not Arabic, will be translated to Arabic (local language), prior to study by 2 translators whose first language is Arabic. Next step, each questionnaire will be translated back to English by a dietitian whose first language is English and who also knows Arabic. All questionnaires will be validated by running them on 10 patients and accordingly modifying their feasibility to the Emirates HD patient's culture, language level and comprehension status.

The physiotherapist and the research assistants will be responsible for training the patients on the exercise program and recording the intensity, duration, and modality of the exercise for each patient as well as patient's complaints and reasons for drop out, if any. The intervention will be given within the HD session: no extra time required beyond the time of HD. During the intervention, patient will be at all times under direct supervision of the physiotherapist and medical team; in case of any discomfort, the intervention will be immediately stopped.

Sample size was chosen based on convenient sampling. Patients of the HD unit who received clearance from the medical team, met the inclusion criteria and consented, were included in the study.

Data will be analyzed through Scientific Package for Social Sciences version 18. Descriptive statistics will be used to analyze the data. Correlations will be conducted through ANOVA. Effect of the study will be analyzed by paired t test on continuous data and Chi-square on categorical data

ELIGIBILITY:
Inclusion Criteria:

* HD patients from the selected HD units in the UAE on HD 3 times a week
* Stable on HD (free of life -threatening acute or chronic disease, with a life expectancy of > 6 months)
* ≥ 3 months on HD
* The gender being irrespective (age ≥ 18)
* Not practicing any physical activity
* With no recent hospitalization (in the last 3 months for ACUTE condition)
* At their full capacity of cognitive, psychiatric and physical ability for self-care and communication
* Capable to communicate either verbally or through writing
* Fully aware of the proposed protocol of the study, and able to provide a consent form.
* All selected patients should have received clearance from their nephrologist and cardiologist that they are eligible to start an exercise program

Exclusion Criteria:

* Patients not meeting the inclusion criteria listed above
* Patients not able to perform the exercise program
* Patients who did not receive the clearance of the attending nephrologist of the unit to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Urea Reduction Ratio (URR) (mmol/L) | Baseline (average of the last 6 months), Week #9,14,18,22,27,31, and at 1 year post intervention
  it is blood urea nitrogen taken pre and post a dialysis session

SECONDARY OUTCOMES:
Exercise Behavior questionnaire | at baseline, end of 6 month intervention, and at 1 year post intervention
  questionnaire
Quality of Life | at baseline, end of 6 month intervention, and at 1 year
  EQ-5D-5L questionnaire
Malnutrition- Inflammation Syndrome | at baseline, end of 6 month intervention, and at 1 year post intervention
  questionnaire
Exercise Fitness Level | Week #1,9,14,18,22,27,31
  assessed through both the BORG scale (exertion level measurement) and heart rate (pulse per minute)
Serum Phosphorous (mmol/L) | Baseline (average of the past 6 months), Week #9,14,18,22,27,31, and at 1 year post intervention
  Blood test
β-aminoisobutyric acid (μM) | at baseline and at post 6 month intervention
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: mirey Karavetian, PhD, Principal Investigator — Zayed University
Locations (1):
- AL Qassimi Hospital, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magnard J, Deschamps T, Cornu C, Paris A, Hristea D. Effects of a six-month intradialytic physical ACTIvity program and adequate NUTritional support on protein-energy wasting, physical functioning and quality of life in chronic hemodialysis patients: ACTINUT study protocol for a randomised controlled trial. BMC Nephrol. 2013 Nov 26;14:259. doi: 10.1186/1471-2369-14-259. PMID 24279747
- [Background] Sheng K, Zhang P, Chen L, Cheng J, Wu C, Chen J. Intradialytic exercise in hemodialysis patients: a systematic review and meta-analysis. Am J Nephrol. 2014;40(5):478-90. doi: 10.1159/000368722. Epub 2014 Dec 9. PMID 25504020
- [Background] Heiwe S, Jacobson SH. Exercise training in adults with CKD: a systematic review and meta-analysis. Am J Kidney Dis. 2014 Sep;64(3):383-93. doi: 10.1053/j.ajkd.2014.03.020. Epub 2014 Jun 7. PMID 24913219
- [Background] Mohseni R, Emami Zeydi A, Ilali E, Adib-Hajbaghery M, Makhlough A. The effect of intradialytic aerobic exercise on dialysis efficacy in hemodialysis patients: a randomized controlled trial. Oman Med J. 2013 Sep;28(5):345-9. doi: 10.5001/omj.2013.99. PMID 24044062
- [Background] Fiaccadori E, Sabatino A, Schito F, Angella F, Malagoli M, Tucci M, Cupisti A, Capitanini A, Regolisti G. Barriers to physical activity in chronic hemodialysis patients: a single-center pilot study in an Italian dialysis facility. Kidney Blood Press Res. 2014;39(2-3):169-75. doi: 10.1159/000355793. Epub 2014 Jul 29. PMID 25117942
- [Background] Kalantar-Zadeh K, Kopple JD, Humphreys MH, Block G. Comparing outcome predictability of markers of malnutrition-inflammation complex syndrome in haemodialysis patients. Nephrol Dial Transplant. 2004 Jun;19(6):1507-19. doi: 10.1093/ndt/gfh143. Epub 2004 Apr 6. PMID 15069177
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- See also: McArdle, W.D., Katch, F.L. & Katch, V. Exercise Physiology: Nutrition, Energy and Human Performance Hardcover - 1 Nov 2009. — http://www.amazon.co.uk/Exercise-Physiology-Nutrition-Performance-William-D-McArdle/dp/1608318591